CLINICAL TRIAL: NCT05080595
Title: Pilot Randomized Controlled Trial of a Need-Based Transportation Assistance Program in Liver Transplant Candidates
Brief Title: Transportation Assistance Program for Liver Transplant
Acronym: TAP-LT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kali Zhou, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-21-00576
Record Dates: First submitted 2021-09-30; First posted 2021-10-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Liver Transplantation
Keywords: transportation; health services; intervention trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transportation assistance, reports unreliable transportation (Experimental): Lyft rides provided to transplant-related appointments
  Interventions: Other: Transportation assistance (Lyft rides)
- No transportation assistance, reports unreliable transportation (No Intervention): No intervention, standard-of-care
- Transportation assistance, control (No Intervention): No intervention, standard-of-care

INTERVENTIONS:
Other: Transportation assistance (Lyft rides) — Lyft rides will be provided to patients for any transplant-related medical visits
  Arms: Transportation assistance, reports unreliable transportation

SUMMARY:
We propose a rideshare-supported intervention that leverages a partnership with Lyft Health, a HIPAA-secured logistics solution that enables us to provide reliable and efficient transportation for patients. Lyft rides will be provided to patients for any transplant-related medical visits, including but not limited to clinic visits with transplant providers, laboratory testing, and imaging/procedural testing that need to be performed as part of the routine evaluation process and prior to waitlisting for transplant.

DETAILED DESCRIPTION:
Transportation barriers are often cited as barriers to healthcare access, leading to delays in care, non-compliance, and lower health outcomes. We hypothesize that access to transportation is a key modifiable social determinant that, if intervened upon, will lead to improvements in equitable access to the liver transplant waitlist (and transplant) for underserved liver transplant candidates.

We propose a rideshare-supported intervention that leverages a partnership with Lyft Health, a HIPAA-secured logistics solution that enables us to provide reliable and efficient transportation for patients. Lyft rides will be provided to patients for any transplant-related medical visits, including but not limited to clinic visits with transplant providers, laboratory testing, and imaging/procedural testing that need to be performed as part of the routine evaluation process and prior to waitlisting for transplant.

Aim 1 is to ascertain the prevalence of transportation barriers among liver transplant candidates and describe the sociodemographic and clinical characteristics of this population. Aim 2 is to pilot a randomized controlled trial of the needs-based app-supported transportation assistance program (TAP-LT) intervention. We will also assess preliminary efficacy, feasibility, patient acceptability, and cost of the intervention. We will conduct a prospective observational survey study (Aim 1) and pilot randomized controlled trial (Aim 2) at a single liver transplant program (Keck Liver Transplant Program at Keck Medical Center).

For the interventional trial, we will have three arms (Figure 2). Participants who report transportation barriers will be randomized 1:1 to either TAP-LT intervention or usual care (no transportation resources or assistance provided). Additionally, participants who report a reliable source of transportation will be included as a secondary control. In this pilot trial, we will enroll 20 participants in each of the three arms. We anticipate initiation of recruitment within 2 months of study approval, recruitment over approximately 6 months, with 6-12 months of intervention and follow-up with the goal of at least 90 days of follow-up after the end of intervention period for all recruited participants. The target population is adult liver transplant candidates who do not have a reliable source of transportation for their healthcare-related visits and needs. We will include adult patients who are eligible for liver transplantation and attend an initial outpatient evaluation visit.

The primary endpoint is the proportion of liver transplant candidates who report barriers to transportation. We will compare sociodemographic and clinical characteristics stratified by transportation status using Chi-square or t-test/Kruskal-Wallis as appropriate. Predictors of transportation barriers will be assessed with univariate and multivariate logistic regression. The primary outcome (time to listing for transplant waitlisting) will be a time-to-event outcome and we will examine the effect of the TAP-LT intervention with intention-to-treat Fine and Gray competing risk regression based on treatment arm. Secondary outcomes will be compared using Chi-square or t-test/Kruskal-Wallis as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+)
* Attended Phase 1 or Phase 1/2 Liver Transplant clinic visit

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant women or prisoners
* Deemed ineligible for liver transplantation during initial evaluation visit
* Not referred for Phase 2 visit at the time of Phase 1 visit among those with initial Phase 1 visit only
* Hospitalized at the time of initial Phase 1 or Phase1/2 visit
* No access to handheld or landline telephone
* Residence outside of 60 miles from Keck Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to waitlisting for liver transplant | through study completion, an average of 1 year
  The primary outcome will be time to waitlisting for liver transplant, defined as time (in days) from initial evaluation visit date to date of official listing for liver transplant in the United Network for Organ Sharing database.

SECONDARY OUTCOMES:
Proportion with reported transportation barriers | 1 year
  Number of patients who report transportation barriers vs those who don't will be obtained from our transportation barriers survey
Proportion waitlisted/transplanted | through study completion, an average of 1 year
  Proportion waitlisted/transplanted will be obtained from medical records
Number of no-shows/cancellations | through study completion, an average of 1 year
  Number of no-shows/cancellations will be obtained from medical records
Number of hospitalizations | through study completion, an average of 1 year
  Number of hospitalizations will be obtained from medical records
Time to transplant | through study completion, an average of 1 year
  Time to transplant will be obtained from medical records
Patient survival at 90 days | through study completion, an average of 1 year
  Vital status will be obtained from medical records
Ride-related data among intervention participants | through study completion, an average of 1 year
  Number of rides, distance/commute time, cost
Patient satisfaction with care | through study completion, an average of 1 year
  Measured by patient satisfaction survey

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Transplant Clinic, Los Angeles, California, United States